CLINICAL TRIAL: NCT06979154
Title: Pilot Study Using Endogenous Aperiodic Brain Activity to Personalize Transcranial Alternating Current Stimulation as a Treatment for Antenatal Depression: PandA-tACS
Brief Title: Pilot Study of Personalized Aperiodic Transcranial Alternating Current Stimulation in Antenatal Depression (PandA-tACS)
Acronym: PandA-tACS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Brain & Behavior Research Foundation (Other); Michigan State University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 25-0425
Record Dates: First submitted 2025-05-08; First posted 2025-05-18 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-08

CONDITIONS: Antenatal Depression; Major Depressive Disorder; Major Depressive Disorder in Pregnancy; Healthy Controls
Keywords: Behavioral Symptoms; Mood Disorders; Mental Disorders; Depression; Depressive Disorder; Major Depressive Disorder; Antenatal diagnoses; Prenatal diagnoses; Pregnancy; Electric Stimulation; non-invasive brain stimulation; transcranial alternating current stimulation; tACS; EEG; antenatal depression; Healthy Controls; Aperiodic brain activity
MeSH Terms: conditions — Depressive Disorder, Major; Behavioral Symptoms; Mood Disorders; Mental Disorders; Depression; Depressive Disorder

STUDY DESIGN:
Intervention Model Description: First phase of study involves healthy controls. Second phase of study involves patients with antenatal depression.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Healthy Control Group (Experimental): Aperiodic tACS delivered using a waveform based on individual participant EEG activity which has been modified to alter excitation/inhibition balance.
  Interventions: Device: tACS (aperiodic)
- Antenatal Depression Group (Experimental): Aperiodic tACS delivered using a waveform based on individual participant EEG activity which has been modified to alter excitation/inhibition balance.
  Interventions: Device: tACS (aperiodic)

INTERVENTIONS:
Device: tACS (aperiodic) — Individualized tACS waveform based on aperiodic EEG activity will be delivered.

SUMMARY:
The purpose of this study is to develop the safety, feasibility, and tolerability of a personalized transcranial alternating current stimulation (tACS) approach in antenatal depression.

DETAILED DESCRIPTION:
The purpose of this study is an initial pilot study to develop the safety, feasibility, and tolerability of a novel, individualized transcranial alternating current stimulation (tACS) approach in antenatal depression, which delivers personalized stimulation waveforms based on the aperiodic component of individual participant EEG activity (PandA-tACS). In Phase I, five healthy controls will receive five consecutive days of PandA-tACS. High-density electroencephalography will be collected at Baseline, D1 and D5, as well as intermittently throughout stimulation sessions. Symptoms will be checked at FUP1 (two weeks following intervention). In Phase II, PandA-tACS will be expanded into five patients with antenatal depression with the same study design. In addition to HD-EEG measurements, depression and related symptoms will be measured at D1, D5 in these patients. Depression and related symptoms will be measured again FUP1 (two weeks following intervention) and FUP2 (4-6 weeks post delivery). Birth outcomes will be recorded within 90 days of expected delivery date as an additional form of safety monitoring.

Primary Aim: To investigate the safety, feasibility, and tolerability of five days of PandA-tACS in healthy controls (Phase I) and in participants with antenatal depression (Phase II).

Exploratory Aim: To investigate aperiodic EEG changes following five days of PandA-tACS in healthy controls and in participants with antenatal depression. Additionally, changes in depression symptoms will be investigated two weeks following PandA-tACS in antenatal depression.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Female aged 18 - 45
* Capacity to understand all relevant risks and potential benefits of the study as determined by study staff (provision of informed consent)
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Low suicide risk (defined for this study as no active suicidal ideation in the past month and no suicide attempts, preparatory actions, or significant non-suicidal self-harm in the previous 2 years). Risk will be assessed utilizing the C-SSRS screen and triage version with further exploration of positive responses.

For healthy control population:

* Use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation, according to NIH Therapeutics Research Program Guidelines.

Additional for antenatal depression population:

* Between weeks 14-32 of viable singleton pregnancy
* Established obstetric care through UNC
* Pre-identified DSM-5 diagnosis of unipolar, non-psychotic MDD which is confirmed by the DIAMOND
* HDRS-17 score ≥14

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

* DSM-5 diagnosis of severe alcohol use disorder (AUD) within the last 12 months, as evidenced by the DIAMOND
* DSM-5 diagnosis of moderate to severe substance use disorder (excluding tobacco) within the last 12 months, as evidenced by the DIAMOND
* Lifetime history of bipolar disorder, as evidenced by DIAMOND
* Schizophrenia spectrum and other psychotic disorders, as evidenced by DIAMOND
* History of autism spectrum disorder
* Initiated any new psychotropic medication in the 6 weeks prior to screening or had a dose change in the preceding 6 weeks
* Initiated a new course of psychotherapy in the 6 weeks preceding screening
* Received any neurostimulation treatment in the 6 weeks preceding screening
* History of seizures (excluding febrile seizures in childhood or Electroconvulsive Therapy (ECT) induced seizures)
* Neurological disorders that would increase risk of participation or present a significant confounder in the opinion of the investigator (for example, dementia, history of stroke, Parkinson's disease, multiple sclerosis, history of traumatic brain injury with prolonged loss of consciousness, ruptured cerebral aneurysm, previous CNS radiation)
* Previously failed to respond to ECT or transcranial magnetic stimulation (TMS)
* Prior brain surgery and/or brain implants
* Implanted medical device that uses electricity
* Currently enrolled in another clinical trial for depression
* Unstable medical disorder or anything that would place the participant at increased risk or preclude the participant's full compliance with or completion of the study, in the opinion of the Investigator

Additional for the healthy control population:

* Current pregnancy or lactation (as determined by urine pregnancy test)
* History of depression, as evidenced by DIAMOND

Additional for the antenatal depression population:

* History of any of the following conditions:

  * Diabetes (gestational or general history)
  * Pre-term delivery (<37 weeks)
  * Eclampsia
  * Pre-eclampsia with severe features
  * Asthma requiring daily medication
  * Chronic hypertension
  * Immune thrombocytopenia (ITP)
  * Hyperthyroidism requiring medication
  * Pre-pregnancy BMI 40 or more
  * In vitro fertilization (IVF)
  * Mullerian anomaly of uterus
  * Organ transplant
  * Prior history of deep vein thrombosis/pulmonary embolism (DVT/PE) or plan for anticoagulation during pregnancy
  * Fetus with autoimmune hydrops
  * Abnormal placenta
* Current pregnancy:

  * HIV/Hep B/Hep C with detectable viral loads
  * Anemia [Hemoglobin under 11.0] upon entry to prenatal care
  * No scheduled prenatal visits by 15 weeks
  * Placenta previa
  * Placenta accreta spectrum (PAS)
  * Pre-eclampsia
  * Gestational diabetes
  * Gestational hypertension
  * Fetus with abnormal chromosomes
  * Cervical length < 2.5 cm
  * Presence of cerclage or vaginal progesterone to decrease chance of pre-term labor
  * Fetal growth restriction
  * Macrosomia
  * Polyhydramnios
  * Oligohydramnios
  * Rupture of membranes
  * Hyperemesis Gravidarum (HEG)
  * Confirmation testing for Tri 13/18/21
  * Congenital anomalies on anatomy ultrasound that do not resolve with follow-up ultrasound
* Other cause of markedly high-risk pregnancy as determined by the Investigator

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Safety via the presence of any serious AEs related to stimulation | Day 1 to Follow-Up (Day 19) (HC) or Day 1 to end of monitoring (birth outcomes review within 90 days of expected delivery date) (antenatal depression)
  The number of serious adverse events reported in healthy control and antenatal depression groups.
Feasibility via the number of participants enrolled relative to the target recruitment in each group | Baseline to end of recruitment period (12 months following recruitment start)
  The number of participants enrolled relative to the target recruitment of five participants in each of the healthy control and antenatal depression groups over the specified 12-month period
Feasibility via the number of participants completing all study visits within the intervention and follow-up period | Healthy controls: Baseline to Follow-Up (Day 19); antenatal depression group: Baseline to Day 5
  The number of participants who complete all study visits within the intervention and follow-up period in the healthy control and antenatal depression groups.
Tolerability via the proportion of participants rating stimulation-related sensations as 'high' | Day 1 to Day 5
  The number of participants who rate stimulation-related sensations as 'high' within the intervention period in the healthy control and antenatal depression groups.
Tolerability via the proportion of participants reporting intolerance to stimulation | Day 1 to Day 5
  The proportion of participants who are unable to tolerate stimulation within the intervention period in the healthy control and antenatal depression groups.
Safety via review of birth outcomes within 90 days of birth in the antenatal depression population | Baseline to end of monitoring (birth outcomes review within 90 days of expected delivery date)
  The number of adverse birth outcomes in participants with antenatal depression. Review will consider length of pregnancy in days, delivery (spontaneous, induced, cesarian (planned or acute), vaginal birth, forceps and/or vacuum extraction), gestational age at birth, Apgar 5 min, malformation, child weight at birth in grams, birth size (small for gestational age, appropriate for gestational age, large for gestational age), neonatal need for intensive care, stillbirth, maternal length of stay in hospital, maternal need for intensive care, pre-eclampsia, as well as EPDS score between 2-4 weeks post-delivery .

OTHER OUTCOMES:
Change in aperiodic exponent following the five-day PandA-tACS intervention | Day 1 to Day 5
  The change in aperiodic exponent from resting state EEG recordings on the first day and the final day of stimulation in healthy control and antenatal depression populations.
Change in HDRS-17 score following intervention in the antenatal depression population | Day 1 up to Follow-up 1 (2 weeks post-stimulation)
  The HDRS-17 is a clinician-administered depression assessment and consists of 17 items with a total score range from 0 to 52. A higher score indicates a worse outcome. Investigators will determine the change in scores across the intervention from Day 1 to Day 5, Day 1 to Follow-up 1, Day 5 to Follow-up 1
Change in Edinburgh Postnatal Depression Scale (EPDS) in the antenatal depression population | Day 1 up to Follow-up 1 (2 weeks post-stimulation)
  The EPDS is a self-administered questionnaire designed to screen for potential symptoms of depression during pregnancy and the postpartum period. This scale consists of 10 short statements, where the participant checks off one of four possible answers about how they have been feeling for the past week. Responses are scored from 0-3, where total scores above 12 or 13 are likely to be suffering from depression. Investigators will determine the change in scores between across the intervention from Day 1 to Day 5, Day 1 to Follow-up 1, Day 5 to Follow-up 1.
Change in Snaith-Hamilton Pleasure Scale (SHAPS) in the antenatal depression population | Day 1 up to Follow-up 1 (2 weeks post-stimulation)
  The SHAPS is a 14-item scale which assesses for anhedonia (the inability to experience pleasure) where each item has a set of four response categories (definitely agree=1, agree=2, disagree=3, definitely disagree=4). Participants are considered to be experiencing mild anhedonia if they disagree with three or more statements. Participants can agree or disagree on a minimum of 0 and maximum of 14 statements. Investigators will determine the change in scores across the intervention from Day 1 to Day 5, Day 1 to Follow-up 1, Day 5 to Follow-up 1.
Change in Clinical Global Impression Scale (CGI) in the antenatal depression population | Day 1 up to Follow-up 1 (2 weeks post-stimulation)
  The CGI is a measure of symptom severity, treatment response and the efficacy of treatments. The CGI involves a single question for the clinician, who rates how mentally ill the participant is, on a scale from 1 (normal), 2 (borderline mentally ill), 3 (mildly ill), 4 (moderately ill), 5 (markedly ill), 6 (severely ill) and 7 (among the most extremely ill participants). Investigators will determine the change in scores across the intervention from Day 1 to Day 5, Day 1 to Follow-up 1, Day 5 to Follow-up 1.
Change in Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q-SF) in the antenatal depression population | Day 1 up to Follow-up 1 (2 weeks post-stimulation)
  The Q-LES-Q-SF is a self-report measure of enjoyment and satisfaction in daily functioning. The total score ranges from 14 to 70, and is expressed as a percentage of the maximum total score that is achievable, where a percentage score ranging from 70-100 is generally indicative of a normal population. Investigators will determine the change in scores across the intervention by comparing scores from Day 1 to Day 5, Day 1 to Follow-up 1, Day 5 to Follow-up 1.
Change in HDRS-17 score following intervention in the antenatal depression population (postnatal period) | Follow-up 1 (2 weeks post-stimulation) to Follow-up 2 (4-6 weeks post delivery)
  The HDRS-17 is a clinician-administered depression assessment and consists of 17 items with a total score range from 0 to 52. A higher score indicates a worse outcome. Investigators will determine the change in scores across the intervention from Follow-up 1 (2 weeks post-stimulation) to Follow-up 2 (4-6 weeks post delivery)
Change in Edinburgh Postnatal Depression Scale (EPDS) in the antenatal depression population (postnatal period) | Follow-up 1 (2 weeks post-stimulation) to Follow-up 2 (4-6 weeks post delivery)
  The EPDS is a self-administered questionnaire designed to screen for potential symptoms of depression during pregnancy and the postpartum period. This scale consists of 10 short statements, where the participant checks off one of four possible answers about how they have been feeling for the past week. Responses are scored from 0-3, where total scores above 12 or 13 are likely to be suffering from depression. Investigators will determine the change in scores between Follow-up 1 (2 weeks post-stimulation) to Follow-up 2 (4-6 weeks post delivery)
Change in Snaith-Hamilton Pleasure Scale (SHAPS) in the antenatal depression population (postnatal period) | Follow-up 1 (2 weeks post-stimulation) to Follow-up 2 (4-6 weeks post delivery)
  The SHAPS is a 14-item scale which assesses for anhedonia (the inability to experience pleasure) where each item has a set of four response categories (definitely agree=1, agree=2, disagree=3, definitely disagree=4). Participants are considered to be experiencing mild anhedonia if they disagree with three or more statements. Participants can agree or disagree on a minimum of 0 and maximum of 14 statements. Investigators will determine the change in scores across the intervention from Follow-up 1 (2 weeks post-stimulation) to Follow-up 2 (4-6 weeks post delivery)
Change in Clinical Global Impression Scale (CGI) in the antenatal depression population (postnatal period) | Follow-up 1 (2 weeks post-stimulation) to Follow-up 2 (4-6 weeks post delivery)
  The CGI is a measure of symptom severity, treatment response and the efficacy of treatments. The CGI involves a single question for the clinician, who rates how mentally ill the participant is, on a scale from 1 (normal), 2 (borderline mentally ill), 3 (mildly ill), 4 (moderately ill), 5 (markedly ill), 6 (severely ill) and 7 (among the most extremely ill participants). Investigators will determine the change in scores across the intervention from Follow-up 1 (2 weeks post-stimulation) to Follow-up 2 (4-6 weeks post delivery)
Change in Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q-SF) in the antenatal depression population (postnatal period) | Follow-up 1 (2 weeks post-stimulation) to Follow-up 2 (4-6 weeks post delivery)
  The Q-LES-Q-SF is a self-report measure of enjoyment and satisfaction in daily functioning. The total score ranges from 14 to 70, and is expressed as a percentage of the maximum total score that is achievable, where a percentage score ranging from 70-100 is generally indicative of a normal population. Investigators will determine the change in scores across the intervention by comparing scores from Follow-up 1 (2 weeks post-stimulation) to Follow-up 2 (4-6 weeks post delivery)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Frohlich, PhD, MSc ETH, MA, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Carolina Center for Neurostimulation, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared in this study due to the small sample size, which may cause participants to become identifiable.

REFERENCES:
- See also: NeuroConn DC-Stimulator MC — https://info.neurocaregroup.com/hubfs/neuroCare_May_2021/pdf/pb_dcsmc_en.pdf